CLINICAL TRIAL: NCT02935244
Title: Advanced Understanding of Staphylococcus Aureus Infections in Europe - Surgical Site Infections
Acronym: ASPIRE-SSI
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Principal Investigator, Jan Kluytmans, MD PhD, UMC Utrecht
Other Study IDs: NL57595.041.16
Record Dates: First submitted 2016-07-20; First posted 2016-10-17 (Estimated); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Staphylococcus Aureus; Surgical Wound Infection
Keywords: Epidemiology; Staphylococcus aureus; Prospective observational; Surgical site or wound infection
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection; Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * A preoperative blood sample
  * An additional blood sample after an SSI episode
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ASPIRE-SSI is a prospective, observational, multicentre cohort study among adult surgical patients, which aims to determine the incidence of healthcare-associated S. aureus infections, particularly S. aureus surgical site infections (SSIs), across Europe and to assess the most important risk factors for this type of infection.

DETAILED DESCRIPTION:
The primary objective of ASPIRE-SSI is to determine the incidence of S. aureus infections, particularly S. aureus SSIs, in various adult surgical patient populations, and to identify the patient-related, pathogen-related, and contextual risk factors for the development of S. aureus SSI. Using this information, a SSI prediction tool will be derived for future clinical trials and public health interventions aimed at SSI prevention. Furthermore, immunologic features protective against S. aureus SSI will also be assessed.

The knowledge obtained by this study will enable identification of the surgical patients most at risk of developing S. aureus infections, particularly S. aureus SSI, and who would probably benefit most from new interventions given prophylactically and specifically to prevent S. aureus infections.

ELIGIBILITY:
Inclusion Criteria:

* The subject is 18 years of age or older.
* The subject is undergoing 1 of the protocol-defined surgical procedures. The surgical procedure is planned or unplanned.
* The subject has been screened for S. aureus colonization from three body regions: nose, throat, and perineum within 30 days prior to surgery, and based on the preoperative S. aureus colonization status of the subject, the subject qualifies for enrolment in the study cohort.
* Written informed consent has been obtained prior to enrollment in the study cohort.

Exclusion criteria:

* Parallel participation in any experimental study of an anti-Staphylococcus preventive intervention.
* An active diagnosis of a SSI as the reason for surgery.
* Not able to comply with study procedures and follow-up based on Investigator judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing 1 of the protocol-defined surgical procedures are eligible for inclusion in the study. However, enrolment in the study cohort population will be based on preoperative S. aureus colonization. In total, approximately 3300 S. aureus colonized subjects and 1700 non-colonized subjects will be enrolled in the study cohort population.
  Protocol-defined surgical procedures: Coronary artery bypass grafting; ICD implantation; knee and hip prosthesis surgery; laminectomy and spinal fusion surgery; emergency surgery; central artery reconstructive and peripheral artery bypass surgery; mastectomy; and craniotomy.
Sampling Method: Non-Probability Sample
Enrollment: 5004 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Incidence of S. aureus SSI | Up to 90 days following surgery.

SECONDARY OUTCOMES:
Incidence of serious S. aureus SSI (deep and organ/space S. aureus SSI) | Up to 90 days following surgery
Incidence of S. aureus bloodstream infection | Up to 90 days following surgery
Incidence of other post-surgical S. aureus infection | Up to 90 days following surgery
Incidence of all-cause SSI, by etiologic agent | Up to 90 days following surgery
Incidence of S. aureus SSI stratified by antibiotic susceptibility | Up to 90 days following surgery
Prevalence of preoperative S. aureus colonization in nose, throat and perineal region. | No more than 30 days prior to surgery
Incidence of S. aureus SSI stratified by location of preoperative S. aureus colonization | Up to 90 days following surgery
Incidence of post-surgical all-cause mortality | Up to 90 days following surgery
Semi-quantification of the bacterial load of colonizing S. aureus | At the time of preoperative screening for S. aureus colonization (within 30 days prior to surgery)
Characterization of S. aureus isolates involved in colonization | At the time of preoperative screening for S. aureus colonization (within 30 days prior to surgery)
  Clonal type, gene sequence, and expression of certain virulence factors of S. aureus isolates
Serum antibody levels against S. aureus virulence factors. | Within 30 days prior to surgery (for the preoperative sample) and 2-6 weeks following the SSI episode (for the post-SSI sample)
Characterization of S. aureus isolates involved in infections | Up to 90 days following surgery
  Clonal type, gene sequence, and expression of certain virulence factors of S. aureus isolates

OTHER OUTCOMES:
Magnitude of healthcare utilization associated with S. aureus SSI in terms of: a. Duration of length of stay (LOS) b. Incidence of readmissions, including re-interventions due to S. aureus SSI c. Duration of LOS during readmissions | Up to 90 days following surgery
Incidence of S. aureus SSI, stratified by participating country | Up to 90 days following surgery
Incidence of S. aureus SSI, stratified by type of surgery | Up to 90 days following surgery
Incidence of S. aureus SSI, stratified by wound classification | Up to 90 days following surgery
Incidence of S. aureus SSI, stratified by urgency of surgery | Up to 90 days following surgery
Incidence of S. aureus SSI, stratified by American Society of Anesthesiologists Physical Score classification | Up to 90 days following surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jan AJW Kluytmans, MD PhD, Principal Investigator — UMC Utrecht
Locations (33):
- Belgium (2):
  - Algemeen Ziekenhuis Sint-Lucas & Volkskliniek Gent, Ghent
  - H. Hartziekenhuis, Lier
- Czechia (4):
  - St. Anne's University Hospital Brno, Brno-střed
  - University Hospital Hradec Kralove, Nový Hradec Králové
  - University Hospital Ostrava, Ostrava
  - University Hospital Motol, Prague
- Estonia (2):
  - North Estonia Medical Centre, Tallinn
  - Tartu University Clinic, Tartu
- Centre Hospitalier Universitaire de Limoges, Limoges, France
- Italy (3):
  - Azienda Ospedaliera Universitaria Ospedali Riuniti, Ancona, Ancona
  - BRESCIA Hospital, Brescia
  - Ospedale Infermi di Rimini, Rimini
- Netherlands (3):
  - Wilhemina Ziekenhuis Assen, Assen
  - Amphia Hospital, Breda
  - UMC Utrecht, Utrecht
- Romania (4):
  - Carol Davila University of Medicine and Pharmacy Bucharest, Bucharest
  - Elias university emergency hospital, Bucharest
  - Prof. C.C. Iliescu Cardiovascular Diseases Institute, Bucharest
  - Clinic County Hospital Timisoara, Timișoara
- Serbia (3):
  - Clinical Centre of Serbia, Belgrade
  - Institute for Orthopedic Surgery Banjica, Belgrade
  - Clinical Centre of Kragujevac, Kragujevac
- Spain (5):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Universitari del Mar, Cadiz
  - HU Reina Sophia, Córdoba
  - Hospital Universitario Central de Asturias, Oviedo
  - Hospital Universitario Virgen Macarena, Seville
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Brighton & Sussex University Hospital NHS Trust, Brighton
  - Derby Teaching Hospitals NHS Foundation Trust, Derby
  - The Pennine Acute Hospitals NHS Trust Manchester, Manchester
  - South Tees Hospitals NHS Foundation Trust, Middlesbrough
  - York Teaching Hospitals NHS Foundation Trust, York

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Design paper — https://www.medrxiv.org/content/10.1101/2020.07.08.20148791v1